CLINICAL TRIAL: NCT00311285
Title: Physical and Mental Load During Laparoscopic Tasks. A Prospective Randomized Trial of the Ergonomics in a Black Box Model
Brief Title: Physical and Mental Load in the Surgeon Performing Laparoscopic Tasks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: BB-001-G-2006
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2006-03

CONDITIONS: Stress
Keywords: Electromyography; Glucocorticoids; Heart Rate; Physical workload; Mental workload; Ergonomics; Laparoscopy; Workload; Biomechanics
MeSH Terms: interventions — Electromyography

INTERVENTIONS:
Device: Electrogram (EMG), heart rate variability (HRV), salivary cortisol, goniometry, inclinometry

SUMMARY:
The surgeons load during laparoscopic surgery is still unclear. Laparoscopic surgery is more demanding because of the challenge of operating through small scars in the abdominal wall without any tactile feedback depending only on the visual feedback on a monitor. The purpose is to establish a model of how to measure mental and physical load in laparoscopy.

DETAILED DESCRIPTION:
The surgeons load during laparoscopic surgery is still unclear. Laparoscopic surgery is more demanding because of the challenge of operating through small scars in the abdominal wall without any tactile feedback depending only on the visual feedback on a monitor. Most studies have been conducted in laboratory set-ups: Black Box.

This study will establish a model of how to measure the biomechanical loads at muscular, joint and postural level, as well as measuring stress-hormone and cardiac rhythm. The study is a precursor of ergonomic studies performed inside the operating room. Advanced operating rooms designed specially for laparoscopy have been introduced in many departments. We do not know if they are more ergonomically correct. We will simulate laparoscopic tasks in an operating room. The hypothesis is that a traditional laparoscopic set-up is more demanding than a set-up mimicking an advanced operating room.

ELIGIBILITY:
Inclusion Criteria:

* Healthy doctors

Exclusion Criteria:

* Pregnancy
* Left handed
* Endocrine disease
* Cardiac rhythm disturbances
* History of recent injury in shoulder/arms

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Study Completion 2007-03

PRIMARY OUTCOMES:
EMG
Goniometry
Inclinometry
HRV
Salivary Cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Helga R Munch-Petersen, MD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- UHGentofte, Hellerup, Denmark